CLINICAL TRIAL: NCT00236106
Title: Short Term Growth in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children´s Clinic, Randers (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: BKR-AD-04
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

INTERVENTIONS:
Drug: tacrolimus ointment 0.1%
Drug: mometasone furoate 0.1%

SUMMARY:
Main objective:to assess short term growth in children with atopic dermatitis during treatment with tacrolimus 0.1% and mometasone furoate 0.1%. A singl blind randomised cross over trial including 20 children. The study consists of 5 periods: run in, treatment(1),wash out, treatment(2) and run out. Each period 14 days where the children will use tacrolimus ointment tvice daily, mometasone furoate once daily or moisturizer (in run in wash out and run out)

ELIGIBILITY:
Inclusion Criteria: age 5-14, atopic dermatitis, normal current growth, Tanner 1, informed consent by the parent or guardian, willing and able to comply with study procedures

Exclusion Criteria: Tanner 2-5, treatment of atopic dermatitis with anti-inflammatory agent within 1 week before the first visit, current asthma or rhinoconjunctivitis that requires treatment with glucocorticoids, endocrine diseases, major surgery within 4 weeks prior to visit 1, fever >39.5 for >3 days

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2005-02; Study Completion 2005-06

PRIMARY OUTCOMES:
short term growth during treatment compared to run in

SECONDARY OUTCOMES:
U-EPX
U-nTX
skin prick test

CONTACTS AND LOCATIONS:
Overall Officials: Ole Wolthers, Principal Investigator — Children's Clinic Randers